CLINICAL TRIAL: NCT01676090
Title: An Epidemiologic, Descriptive and Cross-sectional Study of the IGF-1, IGFBP-3 and ALS Normative Ranges in a Healthy Paediatric Spanish Population, Divided Into Chronological Age, Sex and Pubertal Stage
Brief Title: IGF-1, IGFBP3, ALS Normative Ranges in Healthy Pediatric Spanish Population
Acronym: EDISON
Status: Terminated | Type: Observational
Why Stopped: Participant enrolment was lower than expected
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52800-020
Record Dates: First submitted 2012-08-22; First posted 2012-08-30 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: IGF-1 Deficiency
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the normative ranges of the Insulin-like Growth Factor 1 (IGF-1), Insulin-like growth factor-binding protein 3 (IGFBP-3), Acid-Labile Subunit (ALS) according to age, sex and pubertal stage of a healthy paediatric Spanish population.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex of Caucasian parents
* Age: newborns up to and including 18 years of age
* Length/height, weight and body mass index (BMI) within the mean +/- 2SD (Standard Deviation) and in accordance with the growth charts of the 2010 Spanish cross-sectional growth study (Carrascosa Lezcano et al 2010)
* Signed consent by at least one parent or legal guardian (if subject is ≤18 years) and by subject if ≥12 years

Exclusion Criteria:

* Early or advanced puberty (pubertal signs: between 8 and 9 years old in girls, and between 9 and 10 years old in boys), or delayed puberty (no puberty onset in ≥ 13 year-old girls, and in ≥ 14 year-old boys)
* Chronic diseases including, but not limited to, endocrinologic diseases, chromosomal diseases, chronic diseases of renal, hepatic and/or cardiac aetiology, and tumour processes
* An acute disease during the last two weeks prior to recruitment
* Any clinically significant out-of-range lab value
* Healthy paediatric volunteers who are under medical treatment (contraception permitted)
* A family history of short stature (either parent < P3)
* Children born small for gestational age (birth weight, length, or head circumference < P10)
* Adopted children or conceived through in vitro fertilization ( IVF )
* Subjects who are unwilling or unable in the opinion of the investigator or sponsor to undergo all the study procedures

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy paediatric Spanish population
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
IGF-1 levels according to age, sex and pubertal stage in healthy paediatric volunteers | At the time of participant's single study visit (day 1)

SECONDARY OUTCOMES:
IGFBP-3 levels according to age, sex and pubertal stage in healthy paediatric volunteers | At the time of participant's single study visit (day 1)
ALS levels according to age, sex and pubertal stage in healthy paediatric volunteers | At the time of participant's single study visit (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- Spain (9):
  - Fundación Sant Joan de Deu, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital 12 de Octubre, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Miguel Servet, Zaragoza